CLINICAL TRIAL: NCT04778644
Title: Hippocampal Response to Acute Oral Doses of CBD During an fMRI Memory Task
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Godfrey Pearlson, Founding Director Olin Neuropsychiatry Research Center; Professor Yale University, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: HHC-2020-0367
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: CBD
Keywords: CBD; Memory; MRI

STUDY DESIGN:
Intervention Model Description: All subjects will receive both the study drug and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients with psychosis (Experimental): People who are part of a dimensionally-organized psychosis sample spanning several serious mental illness diagnoses including schizophrenia, schizoaffective disorder, or psychotic bipolar I disorder. Eligible participants will be scheduled for two dose visits where they will receive a 600mg CBD dose on one day and a placebo dose on the other day. Doses will be randomized and double-blind. Doses will be administered via oral gel capsules.
  Interventions: Drug: CBD; Drug: Placebo
- Healthy controls (Experimental): People who do not have a diagnosis of schizophrenia, schizoaffective disorder, or psychotic bipolar I disorder. Eligible participants will be scheduled for two dose visits where they will receive a 600mg CBD dose on one day and a placebo dose on the other day. Doses will be randomized and double-blind. Doses will be administered via oral gel capsules.
  Interventions: Drug: CBD; Drug: Placebo

INTERVENTIONS:
Drug: CBD — Oral gel capsule CBD
  Other Names: CBD Oil; Food grade CBD
Drug: Placebo — Oral gel capsule placebo
  Other Names: Placebo CBD

SUMMARY:
Cannabidiol (CBD) is another cannabis plant derivative for which, like THC, there has been extensive research. Unlike THC however, CBD is non-intoxicating and non-psychedelic. CBD has antipsychotic effects. Logically, if CBD opposes THC effects, it may be a potential antipsychotic treatment. The purpose of this pilot research is to show target engagement of the hippocampus with the study drug (CBD versus placebo) in patients who have been diagnosed with schizophrenia, schizoaffective disorder, or bipolar disorder with psychosis compared to healthy controls.

DETAILED DESCRIPTION:
The investigators conjecture that CBD may act both to modify THC effects and to reduce psychosis symptoms (at least in part) through downstream ECS-related mechanisms, both of which actions converge on the hippocampus, a region rich in CB1 receptors. As such, observing hippocampus activity levels using fMRI can be an effective means of measuring CBD target engagement within this pilot study context. The purpose of this pilot research is to show target engagement of the hippocampus with the study drug cannabidiol (CBD) versus placebo, in BSNIP Biotype 3 compared to Biotypes 1 and 2 and to healthy control subjects, during performance of an fMRI paired associated memory task. Here, investigators will use B-SNIP-based observations in already-characterized B-SNIP subjects, to predict in which individuals CBD engages a theoretically-based brain target. In turn (in future planned studies) such engagement may predict CBD treatment responders. At present, CBD is still an experimental drug for psychosis treatment (although now FDA-approved for treatment of specific types of childhood seizures), but one with a rather benign side-effect profile that could easily be added to ongoing antipsychotic treatment. The purpose of the study is to study response to a single, acute dose of CBD compared to placebo, under double-blind conditions in a small-scale pilot study.

ELIGIBILITY:
Inclusion Criteria:

* 18-50y/o
* Males and females of all races and ethnicities
* Able to provide written informed consent
* Able to read, speak, and understand English
* Meet DSM-IV (SCID-based) criteria for schizophrenia, schizoaffective disorder, bipolar I disorder with psychotic features OR healthy controlled with no diagnosed severe mental illness
* No history of adverse normal baseline values for liver function tests (LFTs)

Exclusion Criteria:

* Strongly left-handed individuals defined as a 60:40 or greater ratio of left to right hand preference (assessed using the Edinburgh Handedness Inventory)
* Premorbid intellectual ability estimate below 70 (WRAT-4, Word Reading subtest, age-corrected standardized score)
* Comorbid DSM-IV diagnosis of alcohol or substance abuse in prior 1 month or substance dependence in prior 3 months
* Neurological (e.g., seizure disorder, stroke, traumatic brain injury with a loss of consciousness ≥ 30min) or severe medical condition (e.g., decompensated cardiovascular disorder, AIDS) that may affect central nervous system function
* Concomitant medications that may interact with study drug adversely such as platelet inhibitors, benzodiazepines, or valproate
* Initial detection of abnormal liver function tests or previous medical history of abnormal liver function or liver disease
* Vulnerable populations (e.g., pregnant, nursing, incarcerated); unwilling to use reliable means of contraception
* High risk for suicide defined as more than 1 attempt in past 12 months that required medical attention, any attempt in the past 3 months or current suicidal ideation with plan and intent such that outpatient care is precluded
* Current homicidal ideation with plan and intent such that outpatient care is precluded
* Positive result on breathalyzer or positive urine toxicology test for any substance, including CBD
* History of prior allergic reaction with CBD or CBD-containing products

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
CBD dose-response for fMRI Hippocampal BOLD values | Post drug administration at 3 hours
  Primary outcome of fMRI-measured hippocampus BOLD values during memory recall task

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey Pearlson, MD, Principal Investigator — Founding Director Olin Research Center; Professor Yale University
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided